CLINICAL TRIAL: NCT03697733
Title: Efficiency of Oral Etoricoxib Versus Intravenous Fentanyl on Post Operative Pain in Curettage Under TIVA : a Randomized Controlled Trial
Brief Title: Comparison Efficiency of Oral Etoricoxib Versus Intravenous Fentanyl on Post Operative Pain in Curettage Under TIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Etovsfen
Record Dates: First submitted 2018-09-28; First posted 2018-10-05 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2018-10

CONDITIONS: Abnormal Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Etoricoxib group (Experimental): Subjects will receive oral Etoricoxib120 mg 30 minutes before fractional curettage then added intravenous Propofol 2 mg/kg when start the procedure
  Interventions: Procedure: fractional curettage
- Intravenous Fentanyl group (Placebo Comparator): Subjects will receive oral placebo [folic acid] 1 tab 30 minutes before the procedure then added intravenous Propofol 2 mg/kg and Intravenous Fentanyl 1 microgram/kg when start the procedure
  Interventions: Procedure: fractional curettage

INTERVENTIONS:
Procedure: fractional curettage — Fractional curettage under TIVA by used oral Etoricoxib120 mg at 30 minutes before fractional curettage and then added intravenous Propofol 2 mg/kg when start the procedure or Intravenous Fentanyl 1 microgram/kg and Propofol 2 mg/kg when start the procedure

SUMMARY:
Comparison of the efficiency of oral Etoricoxib versus intravenous Fentanyl on post operative Pain in curettage under TIVA: A randomized controlled trial

DETAILED DESCRIPTION:
Fractional Curettage is the most widely used for diagnostic and treatment abnormal uterine bleeding. The patient categorize post-operative pain as mild to moderate. Therefore, the effective analgesic added on intraoperative and post-operative is the most important factor in patient's satisfaction, patient well co-operation, shortness time of operation, decrease unpleasant symptoms and rapid recovery. However, there are many anesthetic technique that can be used to relive pain in the operation such as local anesthesia, total intravenous anesthesia, regional anesthesia or oral analgesic drugs.

Intravenous Fentanyl is an short acting opioid. It has a fast onset of action within 2 minutes and short duration of action 30-60 minutes. Respiratory depression, hypotension and bradycardia are adverse effects that might delayed discharge especially in one day surgery e.g. fractional curettage. Etoricoxib is an oral COX-2 specific inhibitor which can be used to relieve the pain. The onset of analgesia can be occurred within 24 minutes which peak plasma level within 60 minutes. There are many empirical evidences to support the results of post-operative pain after used oral Etoricoxib or intravenous Fentanyl. However, there are less evidences to support efficiency of oral Etoricoxib versus intravenous Fentanyl on post-operative Pain in fractional curettage under TIVA

ELIGIBILITY:
Inclusion Criteria:

* Women who having abnormal uterine bleeding undergoing fractional curettage under TIVA

Exclusion Criteria:

* Women who have opioid or NSAIDs allergy
* Women who disagree to participate in this study
* Women who have history of gastrointestinal bleeding or ulcer
* Women who have abnormal kidney function
* Women who can't understand Thai language
* Women who have American Society of Anesthesiologists [ASA] above 2
* Women who have been used NSAIDs in 48 hours or often used NSAIDs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
post operative pain | at 60 minute after operation
  Compare efficacy of oral Etoricoxib and intravenous Fentanyl for post fractional curettage pain by using a visual analog pain scale [Score 0-10]
post operative pain | at 30 minute after operation
  Compare efficacy of oral Etoricoxib and intravenous Fentanyl for post fractional curettage pain by using a visual analog pain scale [Score 0-10]
post operative pain | at 15 minute after operation
  Compare efficacy of oral Etoricoxib and intravenous Fentanyl for post fractional curettage pain by using a visual analog pain scale [Score 0-10]

SECONDARY OUTCOMES:
Adverse effect from the drugs during and post operation | since subject receive drugs until 60 minutes after procedure
  Record subject experience of the following symptoms : nausea and vomiting ,dizziness, drowsiness ,allergic reaction ,chest pain ,and gastrointestinal bleeding or gastrointestinal discomfort
Amount of intravenous Propofol used in the procedure | only intraoperative time
  Record dose of intravenous Propofol that used in TIVA
The first time pain reliever was used in post operation | within 60 minutes after the procedure
  Record the first time patient asked for post operative pain reliver or visual analog pain score > 5

CONTACTS AND LOCATIONS:
Overall Officials: apichaya buraputthananon, Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided